CLINICAL TRIAL: NCT03579888
Title: Donor-Derived Very-Rapid Manufactured CD19-Specific T Cells for Lymphoid Malignancies After Allogeneic Hematopoietic Stem-Cell Transplantation
Brief Title: CD19-Specific T Cells Post AlloSCT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study halted prematurely
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Ziopharm Oncology (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1063; NCI-2020-03608 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1063 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-06-25; First posted 2018-07-09 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: B Acute Lymphoblastic Leukemia With t(v;11q23.3); KMT2A Rearranged; Recurrent B Acute Lymphoblastic Leukemia; Recurrent Chronic Lymphocytic Leukemia; Recurrent Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Recurrent Mantle Cell Lymphoma; Recurrent Non-Hodgkin Lymphoma; Recurrent Ph-Like Acute Lymphoblastic Leukemia; Recurrent Primary Mediastinal (Thymic) Large B-Cell Cell Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory B Acute Lymphoblastic Leukemia; Refractory Chronic Lymphocytic Leukemia; Refractory Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Refractory Mantle Cell Lymphoma; Refractory Non-Hodgkin Lymphoma; Refractory Ph-Like Acute Lymphoblastic Leukemia; Refractory Primary Mediastinal (Thymic) Large B-Cell Cell Lymphoma; Refractory Small Lymphocytic Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (fludarabine, cyclophosphamide, CD19 T cell) (Experimental): CHEMOTHERAPY: Patients receive fludarabine IV over 1 hour and cyclophosphamide IV over 3 hours on days -5, -4, and -3 in the absence of disease progression or unacceptable toxicity.
  T-CELL INFUSION: Patients receive autologous CD19-CD8-CD28-CD3zeta-CAR-mbIL15-HER1t T cells IV over 15-30 minutes on day 0.
  Interventions: Biological: Autologous CD19-CD8-CD28-CD3zeta-CAR-mbIL15-HER1t T Cells; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: Autologous CD19-CD8-CD28-CD3zeta-CAR-mbIL15-HER1t T Cells — Given IV
  Other Names: Autologous CD19-CD8-CD28-CD3zeta-CAR-mbIL15-EGFRt T Cells; CD19-CD8CD28zCAR-specific-mbIL15-HER1t T-lymphocytes
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given IV
  Other Names: Fluradosa

SUMMARY:
This phase I trial investigates the side effects and best dose of CD19 positive (+) specific CAR-T cells in treating patients with CD19+ lymphoid malignancies, such as acute lymphoblastic leukemia, non-Hodgkin lymphoma, small lymphocytic lymphoma, or chronic lymphocytic lymphoma. Sometimes researchers change the genetic material in the cells of a patient's T cells using a process called gene transfer. Researchers then inject the changed T-cells into the patient's body. Receiving the T-cell infusion may help to control the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety and maximum tolerated dose (MTD) of donor-derived genetically modified, CD19-specific T cells expressing mbIL15 and HER1t using the Rapid Personalized Manufacture (RPM) process (autologous CD19-CD8-CD28-CD3zeta-chimeric antigen receptor [CAR]-mbIL15-HER1t T cells [CD19-mbIL15-CAR-T cells]) administered to patients with CD19+ advanced lymphoid malignancies who have previously received an allogeneic hematopoietic stem cell transplantation (HSCT), including haploidentical HSCT.

SECONDARY OBJECTIVES:

I. To demonstrate the feasibility of the RPM process. II. To determine the incidence and grading of cytokine release syndrome (CRS) and neurotoxicity.

III. To determine persistence of genetically modified T cells. IV. To determine if cetuximab can control numbers of infused T cells. V. To screen for the development of host immune responses against the transgenes (one or more of CAR, mbIL15, HER1t).

VI. To determine cytokine profile of the patient with infused T cells. VII. To demonstrate the homing ability of the infused T cells. VIII. To assess disease response after T-cell infusion. IX. To assess progression-free and overall survival. X. To detect emergence of CD19 negative (neg) malignant B cells.

OUTLINE: This is a dose-escalation study of autologous CD19-CD8-CD28-CD3zeta-CAR-mbIL15-HER1t T cells.

CHEMOTHERAPY: Patients receive fludarabine intravenously (IV) over 1 hour and cyclophosphamide IV over 3 hours on days -5, -4, and -3 in the absence of disease progression or unacceptable toxicity.

T-CELL INFUSION: Patients receive autologous CD19-CD8-CD28-CD3zeta-CAR-mbIL15-HER1t T cells IV over 15-30 minutes on day 0.

After completion of study treatment, patients are followed up within 3 days after T-cell infusion and at 1, 2, 3, 4, 6, and 8 weeks, then at 3, 6, and 12 months, then periodically for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* RECIPIENT: Patients with high risk or relapsed disease who are planning to receive, or have received prior allogeneic HSCT from an human leukocyte antigen (HLA)-matched related, or HLA-mismatched related donor; high risk is defined as patients with acute lymphoblastic leukemia who have delayed clearance of minimal residual disease, Philadelphia (Ph)-like, or complex, 11q23 or hypodiploid karyotype
* RECIPIENT: Available donor who provided hematopoietic stem-cell (HSC)
* RECIPIENT: Patients with CD19+ lymphoid malignancies that are refractory to or intolerant of standard treatment (as defined below):

  * B-cell Acute Lymphoblastic Leukemia (ALL)
  * Non-Hodgkin lymphoma (NHL) to include diffuse large B-cell lymphoma (DLBCL) not otherwise specified, primary mediastinal large B cell lymphoma, mantle cell lymphoma, or transformed follicular lymphoma (TFL) as defined by the World Health Organization 2008 criteria
  * Small lymphocytic lymphoma (SLL)
  * Chronic lymphocytic leukemia (CLL)
  * NOTE: Refractory disease for acute and chronic leukemia is defined by:

    * Presence of > 5% malignant blasts in bone marrow and/or peripheral blood and/or minimal residual disease by flow cytometry or molecular analysis for fusion proteins and/or positive imaging for extra-medullary disease to most recent therapy
  * NOTE: Refractory disease for lymphoma is defined as:

    * Progressive disease or stable disease lasting =< 6 months, as best response to most recent chemotherapy regimen; or disease progression or recurrence =< 12 months after prior ASCT
    * Prior therapy must have included an anti-CD20 monoclonal antibody-containing regimen and an anthracycline-containing chemotherapy regimen
    * For patients with TFL, prior chemotherapy for follicular lymphoma and subsequent refractory disease after transformation to DLBCL
    * At least one measurable lesion according to revised International Working Group (IWG) Response Criteria
* RECIPIENT: In patients with prior transplant, treatment will begin no earlier than 3 months post-transplant. Enrollment can occur earlier to allow time for donor cell collection
* RECIPIENT: Karnofsky performance scale > 60
* RECIPIENT: Patient able to provide written informed consent
* RECIPIENT: Patient able to provide written informed consent for the long-term follow-up (LTFU) gene therapy study
* RECIPIENT: Negative human anti-mouse antibody (HAMA)
* DONOR: HLA-matched related, HLA-mismatched related, including haploidentical donor, or related donor cleared to donate based on Stem Cell Transplantation and Cellular Therapy (SCTCT) standard-of-care (SOC) guidelines
* DONOR: Negative beta HCG in female of child-bearing potential defined as:

  * Not post-menopausal for 12 months, or
  * No previous surgical sterilization, or
  * Lactating females
* T-CELL INFUSION REQUIREMENTS FOR RECIPIENT: Patient must have measurable disease at the time of treatment
* T-CELL INFUSION REQUIREMENTS FOR RECIPIENT: Not received anti-thymocyte globulin (ATG), Campath, or other T-cell immunosuppressive antibodies or donor-lymphocyte infusion in the 28 days prior to T-cell infusion
* T-CELL INFUSION REQUIREMENTS FOR RECIPIENT: Serum creatinine < 2 x upper limit of normal (ULN)
* T-CELL INFUSION REQUIREMENTS FOR RECIPIENT: Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) =< 2.5 x ULN or =< 5 x ULN if documented liver metastases
* T-CELL INFUSION REQUIREMENTS FOR RECIPIENT: Total bilirubin =< 1.5 mg/dL, except in patients with Gilbert's syndrome in whom total bilirubin must be =< 3.0 mg/dL
* T-CELL INFUSION REQUIREMENTS FOR RECIPIENT: Cardiac ejection fraction >= 40%, and no clinically-significant electrocardiogram (ECG) findings
* T-CELL INFUSION REQUIREMENTS FOR RECIPIENT: No clinically significant pleural effusion, baseline oxygen saturation > 90% on room air
* T-CELL INFUSION REQUIREMENTS FOR RECIPIENT: No evidence of grade >= 2 active graft versus host disease (GVHD) using the Center for International Blood and Marrow Transplant Research (CIBMTR) Acute GVHD Grading System or requiring systemic steroid therapy greater than physiologic dosing at time of starting treatment
* T-CELL INFUSION REQUIREMENTS FOR RECIPIENT: Non-hematologic toxicity grade >= 2 (Common Terminology Criteria for Adverse Events [CTCAE] version 5) related to the lymphodepleting chemotherapy until the toxicity has resolved to grade =< 1 and the patient is afebrile
* T-CELL INFUSION REQUIREMENTS FOR RECIPIENT: No new grade > 2 neurologic, pulmonary, cardiac, gastrointestinal, renal or hepatic (excluding albumin) toxicity
* T-CELL INFUSION REQUIREMENTS FOR RECIPIENT: Serum creatinine < 2 x ULN
* T-CELL INFUSION REQUIREMENTS FOR RECIPIENT: Oxygen saturation > 90% on room air
* T-CELL INFUSION REQUIREMENTS FOR RECIPIENT: Active clinically significant infection within 7-days of study treatment
* T-CELL INFUSION REQUIREMENTS FOR RECIPIENT: Using an investigational agent

Exclusion Criteria:

* RECIPIENT: Positive beta human chorionic gonadotropin (HCG) in female of child-bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization or lactating females
* RECIPIENT: Patients with allergy to mouse products or cetuximab
* RECIPIENT: Active central nervous system (CNS) disease in patient with history of CNS malignancy
* RECIPIENT: Positive serology for human immunodeficiency virus (HIV)
* RECIPIENT: Active hepatitis B or active hepatitis C
* RECIPIENT: Has received a T-cell product within 6 weeks prior to planned infusion of genetically modified T cells

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 15 years
  Graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Adverse events will be summarized by frequencies and percentages by dose level.
Maximum tolerated dose (MTD) as determined by dose limiting toxicity (DLT) | Up to 30 days post-infusion
  The MTD is defined as the highest dose at which no more than 1 of 6 patients experiences a DLT. The study will employ a standard 3+3 design to find the MTD of CD19-specific chimeric antigen receptor (CAR) T cell dose.

SECONDARY OUTCOMES:
Incidence and grading of cytokine release syndrome (CRS) | Up to 12 months
  Graded according to CTCAE.
Persistence of genetically modified T cells | Up to 12 months
  Persistence of genetically modified T cells will be assessed by the frequency of patients with any detectable CAR-T cells.
Change in numbers of infused T cells | Up to 12 months
  For patients receiving cetuximab (i.e., those who experience >= grade 3 CRS), the change in infused CAR+ T cells from before cetuximab treatment to the nadir of CAR+ T cells after cetuximab summarized by mean, standard deviation, median, and range and days to achieve nadir.
Development of host immune responses against transgenes | Up to 12 months
  The development of host immune responses against the transgenes (one or more of CAR, mbIL15, HER1t) may be assessed by the percentage of patients with antibody formation against each one of the transgenes.
Cytokine levels | Up to 12 months
  Individual patient and aggregate cytokine levels (e.g., IL-15, IL-12, IL-8, etc.) will be summarized by means, standard deviations, medians, and ranges.
Homing ability of the infused T cells | Up to 12 months
  Homing will be assessed based on presence of infused T cells within biopsied tissue. The frequency and percentage of patients experiencing homing and those who have CD19- malignant B cells will be presented.
Disease response | At days 30 and 100
  Percentage of patients experiencing disease response, defined as partial or complete clearance of disease e.g., by positron emission tomography (PET) and/or bone marrow report will be computed along with a corresponding 95% confidence interval. The percentage of patients who had T cells successfully prepared, released, and infused will be reported. Additional statistical analyses will be performed if deemed appropriate.
Neurotoxicity | Up to 12 months
  Graded according to CTCAE.
Presence of CD19 negative (-) malignant B cells | Up to 12 months
  Presence of CD19- malignant B cells will be based on flow cytometry staining for CD19 in the context of staining for antigens to detect cancerous B cells. The frequency and percentage of patients experiencing homing and those who have CD19- malignant B cells will be presented.
Progression-free survival | From the time of T-cell infusion to date of progression of date of death, assessed up to 12 months
  Will be estimated using the Kaplan-Meier method and presented along with their 95% confidence intervals. Additional statistical analyses will be performed if deemed appropriate.
Overall survival | From the time of T-cell infusion to date of death, assessed up to 12 months
  Will be estimated using the Kaplan-Meier method and presented along with their 95% confidence intervals. Additional statistical analyses will be performed if deemed appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Partow Kebriaei, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org